CLINICAL TRIAL: NCT00347503
Title: Aqueous Concentrations and PGE2 Inhibition of Ketorolac 0.4% vs. Bromfenac 0.09% in Cataract Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2601
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2007-07-13 (Estimated); Status verified 2007-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Ketorolac

INTERVENTIONS:
Drug: ketorolac 0.4%, bromfenac 0.09%

SUMMARY:
Evaluation of the aqueous concentrations of 2 topical NSAIDS as well as the PGE2 inhibition in human patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male/Female 21 years of age of older.
* Patient understands and is willing to sign the written informed consent form
* Likely to complete the entire course of the study.
* Patient is scheduled to undergo cataract surgery
* Female patients of childbearing potential must have had a regular menstrual cycle prior to study entry (a female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation).
* Patient is willing and able to administer eye drops and record the times the drops were instilled

Exclusion Criteria:

* Patient has been using a topical NSAID within 1 week of study entry
* Patient has a known sensitivity to any of the ingredients in the study medications
* Patient has sight in only one eye
* Patient has a history of previous intraocular surgery
* Patient's doctor has determined they have a condition (i.e., UNCONTROLLED systemic disease) or are in a situation that may put them at significant risk, confound the study results or may interfere significantly with their participation in the study
* Female patients who are pregnant, nursing an infant or planning a pregnancy
* Patients who are currently involved in another investigational study or have participated in one within the 30 days prior to entering this study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Frank Bucci, Principal Investigator — Bucci Vision Center
Locations (1):
- Bucci Laser Vision, Wilkes-Barre, Pennsylvania, United States